CLINICAL TRIAL: NCT03871426
Title: Manual Cervical Traction and Trunk Stabilization Causes Significant Changes in Lower and Upper Esophageal Sphincter
Brief Title: Manual Therapy Effects on Upper and Lower Esophageal Sphincter Pressures
Status: Completed | Type: Observational
Sponsor: University Hospital, Motol (Other)
Responsible Party: Principal Investigator, Alena Kobesova, Clinical Professor, University Hospital, Motol
Other Study IDs: GERD2_2019
Record Dates: First submitted 2019-03-08; First posted 2019-03-12 (Actual); Last update posted 2019-06-14 (Actual); Status verified 2019-06

CONDITIONS: Gastroesophageal Reflux Disease; Globus Pharyngeus
Keywords: High resolution manometry; globus pharyngeus; gastroesophageal reflux disease; manual cervical traction; trunk stabilization maneuver
MeSH Terms: conditions — Gastroesophageal Reflux; Globus Sensation | interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: manual therapy — Manual Cervical Traction, Trunk Stabilization Maneuver

SUMMARY:
The aim of this study is to test the influence of manual cervical traction and chest stabilization maneuvers on pressures in upper and lower esophageal sphincters.

DETAILED DESCRIPTION:
High Resolution Manometry (HRM) will be used to measure pressure changes in upper esophageal sphincter (UES) and lower esophageal sphincter (LES) during manual cervical traction and trunk stabilization maneuvers. 50-55 gastroesophageal reflux disease (GERD) subjects will participate in the study. UES and pressures will first be measured in relaxed supine position then, during manual cervical traction and finally, the subjects will undergo manual positioning of the trunk into neutral position and LES and UES pressures will be measured again.

ELIGIBILITY:
Inclusion Criteria:

* Gastroesophageal reflux disease

Exclusion Criteria:

* Previous gastro- esophageal surgery
* Concomitant other chronic disease that would affect esophageal motility
* Esophageal structural pathology
* Massive hiatus hernia

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Gastroesophageal reflux disease
Sampling Method: Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2019-03-18 (Actual); Primary Completion 2019-06-13 (Actual); Study Completion 2019-06-13 (Actual)

PRIMARY OUTCOMES:
Pressure in upper and lower esophageal sphincter | up to 6 months
  Pressure in upper and lower esophageal sphincter at rest, during cervical manual traction, and during trunk stabilization maneuver

CONTACTS AND LOCATIONS:
Overall Officials: Alena Kobesova, MD, PhD, Principal Investigator — Department of Rehabilitation and Sports Medicine, University Hospital Motol, Prague, Czech Republic
Locations (1):
- Department of Rehabilitation and Sports Medicine, University Hospital Motol, Prague, Czech Republic, Prague, Czechia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bitnar P, Stovicek J, Andel R, Arlt J, Arltova M, Smejkal M, Kolar P, Kobesova A. Leg raise increases pressure in lower and upper esophageal sphincter among patients with gastroesophageal reflux disease. J Bodyw Mov Ther. 2016 Jul;20(3):518-24. doi: 10.1016/j.jbmt.2015.12.002. Epub 2015 Dec 17. PMID 27634073